CLINICAL TRIAL: NCT01846598
Title: Comparison of 48 Hours After Surgery That Shower and Non-shower Patient's Wound Infection Rate, Pain Score, Patient Satisfaction and Cost.
Brief Title: 48 Hours After Surgery Shower Patient's Wound Infection Rate, Pain Score, Patient Satisfaction and Cost.
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201301038RIND
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Surgical Wound Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
Background and Purpose:The level of the surgical wound healing of the epidermis takes 6-12 hours, and the peak period of 48 hours to achieve healing.The traditional postoperative wound care was every 1-3 days clean with saline and gauze or other dressing and not opened .In traditional concept the wound touch the water that will increase the rate of wound infection.England Department of Health in 2008 surgical wound care guidelines about surgery wound cleaning solution comparison. It was no significant difference in wound infection.with normalsaline and tap water. 2012 The Cochrane Collaboration: Water for wound cleansing systematic review of the literature that wound clean water has no effect on the rate of wound infection and healing rate, conducive to personal hygiene and cost-effective. Under high temperature and humid environments in our country, after surgery not bathe often affect patients' satisfaction and increase the cost of dressing and manpower, Was opened a line after surgery the wound can be shower? It is important about surgical wound care guidelines, but also the patient daily asked a high degree of issues. Purpose of this study (1) post-operative 48 hours, shower or not wound infection rate (2) post-operative 48 hours, shower or not the pain score (3) post-operative 48 hours, shower or not the comfortable (4) post-operative 48 hours, shower or not the care costs.

DETAILED DESCRIPTION:
Methods: In this study, adult patients postoperative 48 hours suture not opened the line and remove the drainage tube of the wound (clean or clean contaminated wounds; the wound category 1,2), single-blind randomized control study. Hospital Research Ethics Committee reviewed and approved, it is expected enrolled 102/04/22-102/12/30, a total of 444 cases, obtained in all cases informed consent form before operation, the case from the hospital Thoracic Surgery, General Surgery , thyroid surgery and orthopedic wards, outpatient closing the case.

Research situations and objects: the subjects conditions: adult (minimum age> 20 years; maximum age are not limit) 48 hours after surgery suture not opened the line and remove the drainage tube wound, closing the case exclusion conditions include: surgical procedure contamination or have been infected wounds, chronic wounds, burns,wounds, trauma wounds, immune function insufficiency or use of immunosuppressive agents can not sign a consent form by the end of the severe and pregnancy.

Research steps: meet the requirements of the subjects to obtain informed consent, by the number of computer random number table, randomly assigned into the shower group or non-shower group, n = 222, shower group will given leaflets before surgery about the wound care guidelines after surgery, (48 hours after surgery, shower not a bath so that your wounds will not be immersed in water, as this may reopen your wounds. please avoid the area of the wound. And gently on your stitches shower, do not vigorously rubbing the wound because it may cause pain,and might delayed wound healing after a rubbing, then with a clean towel and gently pat dry the wound.It can also be allowed to naturally dry or cool air from a hair dryer to dry, do no cover any dressing and maintain open and dry, do not use sanitizer. If shower during hospitalization advised and instructed by researchers. If shower during home, researchers advised and instructed by telephone interviews.The tap water single-use only, unlimited shower time and water amount. Non-shower group were given the current wound care guidance after surgery by the researchers before surgery (without dressing, after 48 hours use sterile normal saline solution clean the wound and cover with gauze, two days to be replaced once, but if sweating or other wet wound, can be replaced at any time.). All subjects returned to the clinic after 7-14 days, the researcher who do not know group will do the wound bacterial culture (if the wound appear red, swelling, heat, pain or purulent exudate or the original physician to determine the need),and the researcher also do outpatient surgical wound photographic archive for all subjects, photographic archive will be sent to an unknown group, MD, Department of Infectious Diseases to determine wound infection (1) or (2) or (3 ): (1) red, swelling, heat, pain (2) purulent exudate (3) bacterial culture (+) the wound track track record with experts validity postoperative.The collected data will Including basic information, the surgical site, surgical start and end times, the use of antibiotics situation, shower time, frequency, cost of water, pain conditions, Comfort, uncomfortable symptoms, surgical wound infection status assessment (skin around the wound redness, swelling, heat, pain, wound pus, exudate type and culture results), wound care costs and frequency. The version SPSS15.0 statistical software for archiving, and T-test ANOVA variance analysis, linear correlation analysis to analyze the data. Outcome measures: wound infection, pain condition, comfort, cost analysis.

ELIGIBILITY:
Inclusion Criteria:

* adult (minimum age> 20 years; maximum age are not limit) postoperative 48 hours suture not opened the line and remove the drainage tube of the wound (clean or clean contaminated wounds; the wound category 1,2)

Exclusion Criteria:

1. surgical procedure contamination or have been infected wounds
2. chronic wounds
3. burns,wounds
4. trauma wounds
5. immune function insufficiency or use of immunosuppressive agents
6. can not sign a consent form
7. the end stage of disease
8. pregnancy

Min Age: 241 Months | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult (minimum age> 20 years; maximum age are not limit) postoperative 48 hours suture not opened the line and remove the drainage tube of the wound (clean or clean contaminated wounds; the wound category 1,2)
Sampling Method: Probability Sample
Enrollment: 444 (Actual)
Dates: Start 2013-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
SURGICAL SITE INFECTION | 7-14 DAYS

CONTACTS AND LOCATIONS:
Overall Officials: Hsieh Pei-Yin, MSD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Fernandez R, Green HL, Griffiths R, Atkinson RA, Ellwood LJ. Water for wound cleansing. Cochrane Database Syst Rev. 2022 Sep 14;9(9):CD003861. doi: 10.1002/14651858.CD003861.pub4. PMID 36103365